CLINICAL TRIAL: NCT07227909
Title: NeuroGuard: Psilocybin Trial for Preventing Chemo-induced Neuropathy
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Usona Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025-1361; NCI-CTRP Clinical Registry (Other: NCI-2025-08499)
Record Dates: First submitted 2025-11-12; First posted 2025-11-13 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Psilocybin; Neuropathy
MeSH Terms: interventions — Psilocybin; Pharmaceutical Preparations; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm A (Experimental): Two supervised oral doses 1 week apart prior to chemotherapy cycle 1 (Day 7 and Day 14), followed by two monthly supervised doses prior to chemotherapy cycles 2 and 3 (Day 42 and Day 70); total 4 doses.
  Interventions: Drug: Psilocybin (drug)
- Arm B (Experimental): Subperceptual dosing every other day for 2 weeks during the pre-chemotherapy run-in (mailed 7×1 mg capsules in tamperevident packaging) prior to the first three cycles as above (21 total doses)
  Interventions: Drug: Psilocybin (drug)
- Arm C (Experimental): Standard of Care: Chemotherapy and supportive care per institutional guidelines; no study drug.
  Interventions: Other: Standard of Care (SOC)

INTERVENTIONS:
Drug: Psilocybin (drug) — Given by po 25 mg
  Arms: Arm A
Drug: Psilocybin (drug) — Given by po 1mg
  Arms: Arm B
Other: Standard of Care (SOC) — No drug
  Arms: Arm C

SUMMARY:
To learn if psilocybin can help to prevent or decrease the severity of chemotherapy-induced peripheral neuropathy (CIPN) in patients who are receiving chemotherapy for the treatment of breast, colorectal, and In this study, psilocybin is being compared to standard supportive care and to a placebo.

DETAILED DESCRIPTION:
Primary Objective

1. To assess the efficacy of psilocybin in the prevention or mitigation of chemotherapy-induced peripheral neuropathy (CIPN) in individuals undergoing adjuvant neurotoxic chemotherapy (i.e., taxanes, platinum-based compounds) for breast, colorectal, and head & neck cancers. The primary endpoint is the proportion of participants with a ≥25% increase (worsening) from baseline to Week 12 on the EORTC QLQ-CIPN20 sensory subscale.

The primary comparison is 25 mg psilocybin vs pooled control (standard of care + 1 mg subperceptual psilocybin), tested two-sided at α=0.05. If significant, two confirmatory pairwise tests (25 mg vs SOC; 25 mg vs 1 mg) will be performed with Hochberg multiplicity control.

Hypothesis: Prophylactic psilocybin administered in four doses (two pre-chemotherapy and two during chemotherapy) will reduce the severity of CIPN as measured by the proportion of participants reporting a 25% or greater increase in CIPN on the EORTC QLQ-CIPN20 sensory subscale compared to placebo or SOC.

Secondary Objectives

1. Determine whether prophylactic psilocybin reduces rates of dose-liming modifications to chemotherapy as result of peripheral neurotoxicity. Dose modifications are defined by either a change in frequency or reduced chemotherapy dose during the 12-week study period. Dose modification decisions will be made by the participant's independent, primary clinician.
2. Determine whether prophylactic psilocybin decreases incidence and severity of CIPN as measured by the NCI-CTCAE criteria
3. Determine whether psilocybin-assisted psychotherapy improves measures of quality of life (e.g., sleep, pain, fatigue, functional status) and psychosocial well-being (e.g., mental health, finding meaning, and post-traumatic growth), as measured by the following: PROMIS-10, PROMIS-A, PROMIS-D, FACT-Cog, PSQI, BFI, MDASI, MEQ30 (mystical experience), Flourishing scale.
4. Determine whether psilocybin-assisted psychotherapy improves functional status per clinicianrated outcome measures.
5. Assess the effects of psilocybin-assisted psychotherapy on all-cause cancer treatment adherence determined by the likelihood that participants will follow the prescribed treatment (adherence) and continue the treatment for the duration prescribed (persistence) for these maintenance therapies.

ELIGIBILITY:
Eligibility Criteria

1. Participants with histologically or cytologically confirmed breast, colorectal, or head and neck cancer.
2. Scheduled to receive platinum-based chemotherapy or taxanes (e.g., paclitaxel, docetaxel).
3. Age 18 years or older
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
5. No pre-existing peripheral neuropathy greater than Grade 1 as defined by the NCI-CTCAE v5.0.
6. No prior grade 3 AEs on current standard of care cancer treatment regimen
7. Must have no major cognitive impairment and be oriented to person, place, and time (e.g. mini mental exam).
8. Must demonstrate willingness to travel to MD Anderson Cancer center for all treatment and follow-up sessions, as well as consent to complete all evaluation instruments and assessments.
9. Agree to abstain from any nicotine products for at least 8-12 hours prior to psilocybin administration until approximately 12 hours after (or when all post-session questionnaires have been completed, whichever comes earlier).
10. Refrain from any psychoactive drugs (including alcohol) for 48 hours prior to psilocybin sessions and must refrain from psychoactive drugs 12 hours after psilocybin sessions. Must consent to urine drug screen (UDS) which will be given before receiving psilocybin. Participants with positive drug test will be retested (UDS) after 6 weeks and included if the repeated UDS is negative. Participant tested positive for a prescribed substance are eligible. Participant failing on the 2nd test (UDS) will be excluded.
11. Must be free from any regularly scheduled psychotropic (antidepressant/anxiolytic class) medications for a minimum of 2 weeks prior to study. Intermittent or PRN use of short-acting anxiolytics or and anti-nausea medications (e.g., ondansetron) may be permitted as defined below in exclusionary criteria). Ondansetron could be taken but must be stopped at least 24 hours before psilocybin administration.
12. Inhibitors of monoamine oxidase, UGT1A9, 1A10, and aldehyde or alcohol dehydrogenase should be discontinued 5 half-lives prior to active dose of psilocybin.
13. Eligible subjects will have a third-party transportation by a licensed driver (e.g. friend, family or a driver) after the psilocybin session is complete. If a driver is used, a friend or family member must accompany them in the vehicle home
14. Participants should agree to refrain from driving, operating heavy machinery, or engaging in safety-sensitive activities for the remainder of the day following psilocybin administration (for both 25mg or subperceptual 1mg placebo).
15. Fluent in English

Exclusion Criteria

1. History of another primary malignancy, except for:

   1. Malignancy treated with curative intent and no active disease for ≥ 5 years before the first dose of study drug, with low potential risk for recurrence.
   2. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
   3. Adequately treated carcinoma in situ without evidence of disease.
2. Clinically significant suicidality or high risk of completed suicide defined as:

   1. Answer 'Yes' to C-SSRS Suicidal Ideation items 4 or 5 within the last 2 months at Screening or 'since last visit' at Baseline
   2. Report having had any C-SSRS Suicidal Behavior item within the past 12 months at Screening or 'since last visit' at Baseline, as defined by 'Yes' to any of the following on the C-SSRS: actual attempt, interrupted attempt, aborted attempt, or preparatory acts
   3. Have any suicidal ideation or thoughts, in the opinion of the study physician or PI, that presents a serious risk of suicidal or self- injurious behavior
3. History of bipolar disorder, psychosis (including a history of schizophrenia).
4. Persons with first-degree relatives who have schizophrenia or other psychotic disorders, or bipolar I or II disorder diagnosed by a qualified mental health professional.
5. Functionally limiting comorbid conditions such as second primary malignancies in CNS or chest, and history of total laryngectomy or total glossectomy precluding them from communicating.
6. ECG with QTc > 450.
7. Participants with non-MRI compatible metal implants.
8. Asymptomatic ALT or AST elevations >/= 5X upper limit of normal, symptomatic ALT or AST elevations >/= 2X upper limit of normal, or total bilirubin >/= 2X upper limit of normal.
9. Uncontrolled diabetes Mellitus with hemoglobin A1c > 8.5%
10. The effects of psilocybin on the developing human fetus are unknown. For this reason, pregnant women will be excluded (Urine test for screening), women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstaining from intercourse with the opposite sex) prior to study entry and for the duration of study participation. This includes all female participants, between the onset of menses (as early as 8 years of age) and 55 years unless the participant presents with an applicable exclusionary factor which may be one of the following:

    * Postmenopausal (no menses in greater than or equal to 12 consecutive months).
    * History of hysterectomy or bilateral salpingo-oophorectomy.
    * Ovarian failure (Follicle Stimulating Hormone and Estradiol in menopausal range, who have received Whole Pelvic Radiation Therapy).
    * History of bilateral tubal ligation or another surgical sterilization procedure.

    Approved methods of birth control are as follows: Hormonal contraception (i.e. birth control pills, injection, implant, transdermal patch, vaginal ring), Intrauterine device (IUD), Tubal Ligation or hysterectomy, Subject/Partner post vasectomy, Implantable or injectable contraceptives, and condoms plus spermicide. Not engaging in sexual activity for the total duration of the trial and the drug washout period is an acceptable practice; however periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
11. Vulnerable populations, including children and cognitively impaired participants, will not be enrolled in this study.
12. Participants with brain metastases.
13. Risk for hypertensive crisis defined as Screening, Baseline, and Medication Session (day of dosing, prior to dosing) blood pressure >180/120mmHG, HR >110 bpm. Of note, we will repeat vital signs for subjects with high initial reading and average three readings to determine eligibility criteria in such cases to account for normal variability in vital sign and "white coat hypertension."
14. Unstable medical conditions or serious abnormalities of complete blood count, chemistries, or ECG that in the opinion of the study physician would preclude safe participation in the trial.

    Some examples include:
    1. Uncompensated congestive heart failure
    2. Clinically significant arrhythmias (e.g., ventricular fibrillation, torsades) or clinically significant ECG abnormality (i.e., QTC interval > 450)
    3. Recent acute myocardial infarction or evidence of ischemia
    4. Malignant hypertension
    5. Congenital long QT syndrome
    6. Acute renal failure
    7. Severe hepatic impairment
    8. Respiratory failure
15. Significant central nervous system (CNS) pathology. Some examples include:

    1. Primary or secondary cerebral neoplasm on imaging
    2. Epilepsy and any history of seizure (regardless of if related to epilepsy) except for a onetime febrile seizure in childhood
    3. History of stroke in the past 3 years
    4. Untreated cerebral aneurysm
    5. Dementia
    6. Ongoing delirium of any kind (including with or without psychosis) in which subjects would not have the capacity to participate in the study.
16. High risk of adverse emotional or behavioral reaction based on investigator's clinical evaluation.

    Examples include:
    1. Agitation
    2. Violent behavior
17. Active substance use disorders (SUDs) defined as: DSM-5 criteria for moderate or severe alcohol or drug use disorder (excluding caffeine and nicotine) within the past year

    a. Extensive use of serotonergic hallucinogens (e.g., LSD, psilocybin) defined as: i. Any use in the last 12 months ii. >22 lifetime uses iii. History of diagnosed hallucinogen persisting perception disorder (HPPD)
18. Concurrent Medications

    1. Antidepressants
    2. Centrally-acting serotonergic agents (e.g., MAO inhibitors)
    3. Antipsychotics (e.g., first and second generation)
    4. Mood stabilizers (e.g., lithium, valproic acid)
    5. Aldehyde dehydrogenase inhibitors (e.g., disulfiram)
    6. Significant inhibitors of UGT 1A0 or UGT 1A10
    7. serotonin-acting dietary supplements (such as 5-hydroxytryptophan or St. John's wort)
    8. efavirenz
    9. Other Medications Listed in Section 3.1 19. Have a positive urine drug test including Amphetamines, Barbiturates, Buprenorphine, Benzodiazepines, Cocaine, Cannabis, Methamphetamine, MDMA, Methadone, Opiates (Morphine, Oxycodone), Phencyclidine (PCP), and Tetrahydrocannabinol (THC).

    <!-- -->

    1. Note: Prescribed opiate medications (e.g., cancer-related pain) will be allowed to continue through the study period for participants who have been on a stable dose of such medicine for at least 1 month prior to Screening, as determined during review of concomitant medications.
    2. Note: Prescribed benzodiazepine medications and nonbenzodiazepine sleeping medications will be allowed to continue through the study period for participants who have been on a stable dose of such a medicine for at least 6 weeks prior to Screening, as determined during review of concomitant medications.
    3. Note: Participants using cannabis, including legal cannabis, for any purposes must agree to refrain from use beginning at Screening, as confirmed with a negative Baseline drug test, and through to the end of the study.
    4. Note: Participants using prescribed psychostimulants (amphetamines and Ritalin), must agree to refrain from use 72 hours prior to dosing and until 12 hours after dosing.

20. Have a psychiatric condition judged to be incompatible with establishment of rapport with the study therapists or safe exposure to psilocybin

1. Have any psychological or physical symptom, medication or other relevant finding prior to randomization, based on the clinical judgment of the PI or relevant clinical study staff that would make a participant unsuitable for the study.
2. Have an allergy or intolerance to any of the materials contained in either drug product Be enrolled in another clinical trial assessing intervention(s) for prevention or treatment of any pain-related symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Estimated)
Dates: Start 2026-05-04 (Estimated); Primary Completion 2029-01-31 (Estimated); Study Completion 2031-01-31 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Moran Amit, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States